CLINICAL TRIAL: NCT04927819
Title: Prospective Observational Study on Evolution of Extra-short Implants (<6.5 mm) Compared to Non-extra-short Implants (≥ 6.5 mm) Splinted on the Same Prosthesis
Brief Title: Extra-short vs. Non-extra-short Dental Implants Splinted on the Same Prosthesis
Status: Recruiting | Type: Observational
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Other Study IDs: FIBEA_02_EP/20/Extracortos
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- short-length implant (<6.5 mm)
  Interventions: Device: BTI Implant
- non-short length implant (≥6.5 mm)
  Interventions: Device: BTI Implant

INTERVENTIONS:
Device: BTI Implant — BTI Dental implants are non-active medical device, single use, non resterilizable, biocompatible and sterile devices made of alloplastic materials (Titanium) intended to be surgically implanted into alveolar and/or basal bone of the mandible or maxilla to provide support and a means of retention for a dental prosthesis (e.g. bridge, single-tooth, overdenture).

SUMMARY:
The main aim of this prospective study is to analyze the survival rate of short-length implants (<6.5 mm) in subjects with partial edentulism. Non-short length implant will be used as control arm. Additionally, others clinical parameters (marginal bone loss and prosthetic associated complications) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Have planned a fixed multiple prosthesis supported by implants <6.5 mm in length and implants ≥ 6.5 mm in length within 15 days before the inclusion of the patient in the study.
* Planning of supported prostheses from 2 to 4 implants dental
* Have a previously performed CBCT (Cone Beam Computed Tomography)
* Availability to be observed during the period of tracing
* Signature of the informed consent

Exclusion Criteria:

* Smokers> 10 cigarettes / day
* Complete prostheses
* Unitary prostheses

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Partial edentulism
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Survival of dental implants | 1 year
  Survival of dental implants at one year post-implantation

SECONDARY OUTCOMES:
Marginal bone loss | 1 year
  Marginal bone loss at one year post-implantation
Incidence of prosthetic or implant complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Anitua, MD, Principal Investigator — Clinica Eduardo Anitua
Locations (1):
- Clinica Eduardo Anitua, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: Undecided